CLINICAL TRIAL: NCT00386009
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multicenter Study to Evaluate the Urodynamic Effects of Tadalafil Once a Day for 12 Weeks in Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: Effects of Tadalafil Once a Day for 12 Weeks in Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11233; H6D-MC-LVHK
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Benign Prostatic Hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): tadalafil
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — 20 mg tadalafil tablet taken by mouth once a day for 12 weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: Placebo — Placebo tablet taken by mouth once a day for 12 weeks.
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the function of the bladder and urethra during urinary storage or voiding in men with signs and symptoms of benign prostatic hyperplasia treated with either placebo or tadalafil.

ELIGIBILITY:
Inclusion Criteria:

* Men 40 years of age or older with Lower Urinary Tract Symptoms (LUTS) with a total International Prostate Symptom Score (IPSS) greater than or equal to 13 at Visit 1.
* Agree not to use any other approved or experimental medications for Benign Prostate Hyperplasia (BPH)-Lower Urinary Tract Symptoms, including alpha blockers, 5-alpha reductase inhibitors, PDE5 inhibitors, or herbal preparations at any time during the study.
* Have not taken finasteride or dutasteride therapy for at least 4 months prior to Visit 2; have not taken any other LUTS therapy (including herbal preparations) or PDE5 inhibitors for at least 4 weeks prior to Visit 2.
* Have had BPH-LUTS for greater than 6 months prior to Visit 1.

Exclusion Criteria:

* Any pelvic surgical procedure on the urinary tract, including minimally invasive BPH-LUTS therapies and penile implant surgery.
* History of urethral obstruction due to stricture, valves, sclerosis, or tumor.
* Current neurologic disease or condition associated with neurogenic bladder (for example, Parkinson's disease, multiple sclerosis).
* History of cardiac conditions including myocardial infarction, bypass surgery, angioplasty or stent placement for a specified time before starting the study.
* History of angina requiring treatment with nitrates.
* Prostate Specific Antigen (PSA) greater than 10 nanogram/milliliter (ng/ml) at Visit 1.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tarzana, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middlebury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Wayne, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden City, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Portugal (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Tadalafil
Started | 101 | 99
Completed | 92 | 89
Not Completed | 9 | 10
Not completed — Adverse Event | 0 | 2
Not completed — Death | 1 | 0
Not completed — Entry Criteria Not Met | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Sponsor Decision | 1 | 1
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil | Total
Number analyzed (Participants) | 101 | 99 | 200
Age Continuous [Mean (Standard Deviation); unit: years] | 59.03 (9.69) | 58.16 (8.82) | 58.60 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 101 | 99 | 200
Region of Enrollment [Number; unit: participants]
  United States | 99 | 95 | 194
  Canada | 2 | 4 | 6
Baseline Benign Prostatic Hyperplasia (BPH) Lower Urinary Tract Symptom (LUTS) Severity [Number; unit: participants] — Severity was determined by the International Prostate Symptom Score (IPSS)Total. The IPSS is obtained by combining the scores of the responses to the 7 component questions. Each question is scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
  participants
    Moderate (IPSS <20) | 34 | 35 | 69
    Severe (IPSS ≥20) | 66 | 62 | 128
    Missing Baseline Measure | 1 | 2 | 3
Bladder Outlet Obstruction Index (BOOI) [Number; unit: participants] — BOOI, or bladder outlet obstruction index, which is derived from the equation: pdetQmax-2Qmax (where pdetQmax is detrusor pressure at peak urinary flow rate and Qmax is defined as the peak urine flow rate).
  participants
    Obstructed (BOOI > 40) | 33 | 34 | 67
    Equivocal (BOOI 20-40) | 35 | 34 | 69
    Unobstructed (BOOI < 20) | 33 | 31 | 64
Duration of Benign Prostatic Hyperplasia Lower Urinary Tract Symptoms (BPH LUTS) [Number; unit: participants]
  6 months to 1 year | 13 | 12 | 25
  1 year to 3 years | 36 | 30 | 66
  > 3 years | 52 | 57 | 109
Erectile Dysfunction Severity [Number; unit: participants] — This measure is only for participants who have Erectile Dysfunction.
  participants
    Mild | 20 | 22 | 42
    Moderate | 31 | 31 | 62
    Severe | 9 | 5 | 14
Presence of Erectile Dysfunction [Number; unit: participants]
  Yes | 60 | 58 | 118
  No | 41 | 41 | 82
Previous Alpha-Blocker Therapy [Number; unit: participants]
  Yes | 22 | 21 | 43
  No | 79 | 78 | 157
Previous Therapy for Benign Prostatic Hyperplasia [Number; unit: participants]
  Yes | 34 | 29 | 63
  No | 67 | 70 | 137
Race/Ethnicity [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 2 | 5
  Black or African American | 12 | 13 | 25
  Hispanic or Latino | 8 | 8 | 16
  White | 78 | 75 | 153
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square centimeters (kg/cm^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square centimeters (kg/cm^2) | 29.44 (4.47) | 29.45 (4.93) | 29.45 (4.69)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 92.94 (16.55) | 93.90 (16.49) | 93.42 (16.49)
Height [Mean (Standard Deviation); unit: centimeters] | 177.56 (8.07) | 178.58 (7.50) | 178.07 (7.79)
Postvoid Residual Volume by Ultrasound [Mean (Standard Deviation); unit: milliliters] | 59.30 (60.87) | 45.65 (49.58) | 52.51 (55.82)
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: nanograms per milliliter] | 1.60 (1.13) | 1.51 (1.14) | 1.55 (1.13)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Week Endpoint in Detrusor Pressure at Peak Urinary Flow Rate (PdetQmax)
Time Frame: Baseline and 12 weeks
Population: Number of participants randomized, had started study medication, had both a baseline and an end-of-study pressure-flow urodynamic assessment, and had at least 37 days (6 weeks minus a 5-day visit window) on treatment between randomization and the final pressure-flow urodynamic assessment.
Measure: Mean (Standard Deviation); unit: centimeters of water (cm H20)
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 91 | 84
centimeters of water (cm H20)
  Baseline | 54.83 (27.36) | 56.87 (29.67)
  Change from Baseline to 12 Week Endpoint | 1.92 (19.71) | -2.95 (15.92)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.068, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

2. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Peak Urinary Flow Rate (Qmax) Measured During Free-Flow Studies
Description: Qmax was measured during free-flow tests using a standard calibrated flow meter.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters per second
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 89 | 82
milliliters per second
  Baseline | 13.03 (7.34) | 14.75 (10.70)
  Change from Baseline to 12 Week Endpoint | 0.52 (7.83) | 0.01 (8.83)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.626, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

3. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Mean Urinary Flow Rate (Qave) Measured During Free-Flow Studies
Description: Qave was measured during free-flow tests using a standard calibrated flow meter.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millilters per second
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 70 | 59
millilters per second
  Baseline | 7.10 (4.37) | 7.23 (4.18)
  Change from Baseline to 12 Week Endpoint | -0.01 (4.11) | 1.00 (3.04)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.113, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

4. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Volume of Voided Urine (Vcomp) Measured During Free-Flow Studies
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 88 | 82
milliliters
  Baseline | 258.56 (134.21) | 268.22 (149.77)
  Change from Baseline to 12 Week Endpoint | -4.10 (151.82) | -5.17 (151.73)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.837, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

5. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Postvoid Residual Volume (PVRcath) Measured During Free-Flow Studies
Description: PVRcath is the volume of urine remaining int he bladder after voiding, measured by catheterization.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 78 | 79
milliliters
  Baseline | 59.62 (66.74) | 48.99 (65.73)
  Change from Baseline to 12 Week Endpoint | -1.85 (80.92) | -9.13 (70.36)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.400, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

6. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Total Bladder Capacity Measured During Free-Flow Studies
Description: Total bladder capacity was defined as Vcomp + PVRcath (obtained when the bladder was full).
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 77 | 78
milliliters
  Baseline | 327.95 (165.66) | 316.79 (187.31)
  Change from Baseline to 12 Week Endpoint | -17.53 (182.62) | -14.88 (187.10)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.864, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

7. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Bladder Voiding Efficiency (BVE) Measured During Free-Flow Studies
Description: Bladder voiding efficiency was defined as (Vcomp/total bladder capacity) X 100 (obtained when the bladder was full).
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 77 | 78
milliliters
  Baseline | 84.01 (14.56) | 85.85 (13.44)
  Change from Baseline to 12 Week Endpoint | -0.52 (16.31) | 1.85 (16.22)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.340, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

8. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Peak Urinary Flow Rate (Qmax) Measured During Pressure-Flow Studies
Description: Qmax was measured duirng pressure-flow tests.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters per second
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 91 | 84
milliliters per second
  Baseline | 9.49 (4.90) | 10.29 (4.46)
  Change from Baseline to 12 Week Endpoint | 0.50 (2.91) | 0.38 (2.92)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.838, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

9. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Mean Urinary Flow Rate (Qave) Measured During Pressure-Flow Studies
Description: Qave was measured during pressure-flow tests.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters per second
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 87 | 81
milliliters per second
  Baseline | 4.67 (2.44) | 5.50 (2.68)
  Change from Baseline to 12 Week Endpoint | 0.45 (1.66) | 0.58 (1.91)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.609, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

10. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Volume of Voided Urine (Vcomp) Measured During Pressure-Flow Studies
Description: Vcomp was defined as the volume of voided urine measured during pressure-flow tests.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 91 | 84
milliliters
  Baseline | 294.10 (147.74) | 296.64 (143.30)
  Change from Baseline to 12 Week Endpoint | 3.31 (140.46) | 13.51 (99.64)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.427, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

11. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Maximum Detrusor Pressure (Max Pdet) Measured During Pressure-Flow Studies
Description: Max Pdet was defined as the maximum detrusor pressure observed during voiding.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters of water (cm H20)
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 83 | 78
centimeters of water (cm H20)
  Baseline | 67.13 (31.66) | 72.20 (38.65)
  Change from Baseline to 12 Week Endpoint | -0.48 (28.19) | -2.11 (24.08)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.838, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

12. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Bladder Contractility Index (BCI) Measured During Pressure-Flow Studies
Description: BCI was derived from the equation PdetQmax + 5Qmax. Scores: <100 means weak, 100-150 menas normal, >150 means strong. A decrease means a decrease in contractility of the bladder.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a nomogram
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 91 | 84
units on a nomogram
  Baseline | 102.28 (32.84) | 108.32 (32.14)
  Change from Baseline to 12 Week Endpoint | 4.43 (20.86) | -1.04 (20.37)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.090, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

13. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Bladder Outlet Obstruction Index (BOOI) Measured During Pressure-Flow Studies
Description: BOOI, formerly known as the Abrams-Griffith number, was derived from the equation PdetQmax - 2Qmax. Scores: <20 means unobstructed, 20-40 means equivocol, >40 means obstructed. An increase means worsening of obstruction, a decreased means lessening of obstruction (improvement).
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a nomogram
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 91 | 84
units on a nomogram
  Baseline | 35.84 (30.87) | 36.28 (33.14)
  Change from Baseline to 12 Week Endpoint | 0.92 (22.10) | -3.71 (17.56)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.113, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

14. Secondary Outcome: Presence of Involuntary Detrusor Contractions During Bladder Filling
Time Frame: Baseline and 12 weeks
Population: Number of participants randomized, had started study medication, had both a baseline and an end of-study pressure-flow urodynamic assessment, and had at least 37 days (6 weeks minus a 5-day visit window) on treatment between randomization and the final pressure-flow urodynamic assessment.
Measure: Number; unit: participants
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 91 | 84
participants
  Present at Baseline | 33 | 28
  Not Present at Baseline | 58 | 56
  Present at Endpoint | 36 | 31
  Not Present at Endpoint | 55 | 53
  Present at Both Baseline and Endpoint | 22 | 18
  Present at Baseline Only | 11 | 10
  Present at Endpoint Only | 14 | 13
  Present at Neither Baseline nor Endpoint | 44 | 43

15. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Bladder Volume at First Involuntary Detrusor Contraction
Description: Assessed in participants with involuntary detrusor contractions during the bladder filling at both baseline and endpoint.
Time Frame: Baseline and 12 weeks
Population: Number of participants in the Primary Analysis Population with involuntary detrusor contractions during bladder filling at both baseline and endpoint.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 22 | 18
milliliters
  Baseline | 120.55 (82.50) | 164.00 (108.31)
  Change from Baseline to 12 Week Endpoint | 27.86 (128.20) | 28.56 (106.67)

16. Secondary Outcome: Change From Baseline to 12 Week Endpoint in International Prostate Symptom Score (IPSS) Total Score
Description: The IPSS Total Score is obtained by combining the scores of the responses to the 7 component questions. Each question is scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 91 | 82
units on a scale
  Baseline | 22.01 (5.72) | 21.46 (5.63)
  Change from Baseline to 12 Week Endpoint | -5.04 (6.93) | -9.13 (6.90)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for Change from Baseline to 12 Week Endpoint. Change = Endpoint minus baseline

17. Secondary Outcome: Clinically Adverse and Statistically Significant Changes From Baseline to 12 Week Endpoint in Laboratory Tests
Description: Laboratory tests that were statistically significant and clinically adverse would be reported for safety.
Time Frame: Baseline and 12 weeks
Population: All randomized participants.
Measure: Number; unit: significant and clinically adverse labs
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 98 | 94
significant and clinically adverse labs | 0 (0.41) | 0 (0.33)

ADVERSE EVENTS:
Arm/Group | Placebo | Tadalafil
Serious Adverse Events (participants affected / at risk) | 2 | 3
Other Adverse Events (participants affected / at risk) | 28 | 55
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Tadalafil
Myocardial infarction/Death (Cardiac disorders) | 1/101 (1) | 0/99 (0)
Cellulitis (Infections and infestations) | 0/101 (0) | 1/99 (1)
Pneumonia (Infections and infestations) | 0/101 (0) | 1/99 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0/101 (0) | 1/99 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0/101 (0) | 1/99 (1)
Hypoaesthesia (Nervous system disorders) | 1/101 (1) | 0/99 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0/101 (0) | 1/99 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Tadalafil
Bradycardia (Cardiac disorders) | 0/101 (0) | 1/99 (1)
Coronary artery disease (Cardiac disorders) | 0/101 (0) | 1/99 (1)
Syncope (Cardiac disorders) | 1/101 (1) | 0/99 (0)
Ear discomfort (Ear and labyrinth disorders) | 0/101 (0) | 1/99 (1)
Vision blurred (Eye disorders) | 0/101 (0) | 1/99 (1)
Visual disturbance (Eye disorders) | 0/101 (0) | 1/99 (1)
Abdominal pain (Gastrointestinal disorders) | 1/101 (1) | 1/99 (1)
Diarrhoea (Gastrointestinal disorders) | 0/101 (0) | 1/99 (1)
Dyspepsia (Gastrointestinal disorders) | 0/101 (0) | 8/99 (8)
Dysphagia (Gastrointestinal disorders) | 0/101 (0) | 1/99 (1)
Flatulence (Gastrointestinal disorders) | 0/101 (0) | 1/99 (1)
Food poisoning (Gastrointestinal disorders) | 0/101 (0) | 1/99 (1)
Gastritis (Gastrointestinal disorders) | 0/101 (0) | 2/99 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0/101 (0) | 3/99 (3)
Haemorrhoids (Gastrointestinal disorders) | 0/101 (0) | 1/99 (1)
Toothache (Gastrointestinal disorders) | 1/101 (1) | 1/99 (1)
Seasonal allergy (Immune system disorders) | 1/101 (1) | 1/99 (1)
Bronchitis (Infections and infestations) | 0/101 (0) | 1/99 (1)
Ear infection (Infections and infestations) | 0/101 (0) | 1/99 (1)
Gastroenteritis aeromonas (Infections and infestations) | 1/101 (1) | 0/99 (0)
Influenza (Infections and infestations) | 1/101 (1) | 2/99 (2)
Nasopharyngitis (Infections and infestations) | 2/101 (2) | 1/99 (1)
Sinusitis (Infections and infestations) | 0/101 (0) | 1/99 (1)
Upper respiratory tract infection (Infections and infestations) | 2/101 (2) | 2/99 (2)
Urinary tract infection (Infections and infestations) | 1/101 (1) | 0/99 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0/101 (0) | 1/99 (1)
Biopsy prostate (Investigations) | 1/101 (1) | 0/99 (0)
Blood creatinine increased (Investigations) | 0/101 (0) | 1/99 (1)
Gamma-glutamyltransferase increased (Investigations) | 0/101 (0) | 1/99 (1)
Hepatic enzyme increased (Investigations) | 0/101 (0) | 2/99 (2)
Liver function test abnormal (Investigations) | 1/101 (1) | 0/99 (0)
Prostatic specific antigen increased (Investigations) | 1/101 (1) | 0/99 (0)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0/101 (0) | 1/99 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/101 (0) | 1/99 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2/101 (2) | 1/99 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1/101 (1) | 0/99 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/101 (0) | 2/99 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1/101 (1) | 0/99 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3/101 (3) | 5/99 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 0/101 (0) | 1/99 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0/101 (0) | 1/99 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1/101 (1) | 0/99 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0/101 (0) | 1/99 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0/101 (0) | 1/99 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0/101 (0) | 1/99 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2/101 (2) | 1/99 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/101 (0) | 2/99 (2)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/101 (1) | 0/99 (0)
Amnesia (Nervous system disorders) | 1/101 (1) | 0/99 (0)
Dizziness (Nervous system disorders) | 3/101 (3) | 0/99 (0)
Headache (Nervous system disorders) | 3/101 (3) | 7/99 (7)
Nerve compression (Nervous system disorders) | 0/101 (0) | 1/99 (1)
Paraesthesia (Nervous system disorders) | 1/101 (1) | 0/99 (0)
Sciatica (Nervous system disorders) | 0/101 (0) | 1/99 (1)
Syncope vasovagal (Nervous system disorders) | 0/101 (0) | 1/99 (1)
Nicotine dependence (Psychiatric disorders) | 1/101 (1) | 0/99 (0)
Dysuria (Renal and urinary disorders) | 0/101 (0) | 1/99 (1)
Haematuria (Renal and urinary disorders) | 1/101 (1) | 1/99 (1)
Urethral pain (Renal and urinary disorders) | 0/101 (0) | 1/99 (1)
Urinary tract disorder (Renal and urinary disorders) | 1/101 (1) | 0/99 (0)
Penis disorder (Reproductive system and breast disorders) | 0/101 (0) | 1/99 (1)
Peyronie's disease (Reproductive system and breast disorders) | 0/101 (0) | 1/99 (1)
Scrotal pain (Reproductive system and breast disorders) | 1/101 (1) | 0/99 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/101 (1) | 0/99 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2/101 (2) | 1/99 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1/101 (1) | 0/99 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/101 (1) | 1/99 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/101 (1) | 0/99 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0/101 (0) | 1/99 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0/101 (0) | 1/99 (1)
Acne (Skin and subcutaneous tissue disorders) | 1/101 (1) | 0/99 (0)
Rash (Skin and subcutaneous tissue disorders) | 0/101 (0) | 2/99 (2)
Cataract operation (Surgical and medical procedures) | 0/101 (0) | 1/99 (1)
Endodontic procedure (Surgical and medical procedures) | 1/101 (1) | 0/99 (0)
Foot operation (Surgical and medical procedures) | 0/101 (0) | 1/99 (1)
Tooth repair (Surgical and medical procedures) | 1/101 (1) | 0/99 (0)
Aortic aneurysm (Vascular disorders) | 0/101 (0) | 1/99 (1)
Flushing (Vascular disorders) | 0/101 (0) | 1/99 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days